CLINICAL TRIAL: NCT00277901
Title: MRI Assessment of Two Congenital Heart Disease States: Assessment of Right Ventricular Function: Predictor of Optimal Timing of Pulmonary Valve Replacement in Patients With TOF; Assessment of Flow Dynamics in Patients With Aortic Coarctation
Brief Title: MRI Assessment of RV Function: Patients With TOF or Aortic Coarctation
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: James Parks, MD, Children's Healthcare of Atlanta Institutional Review Board
Other Study IDs: 02-122
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Congenital Disorders
Keywords: cardiac; pediatric; MRI; Tetralogy of Fallot TOF; Aortic Coarctation
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Aortic Coarctation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
At Children's Healthcare of Atlanta at Egleston, it is standard of care to do a cardiac MRI on patients with the diagnosis of Tetralogy of Fallot and Aortic Coarctation to evaluate heart function. We propose to do a retrospective chart review of patient data along with their MRI data to analyze ventricular function and cavity volumes pre-Tetralogy of Fallot repair, post-Tetralogy of Fallot repair (pre-valve repair/replacement) and post-valve repair/replacement in order to assess the efficacy and optimal timing of valve replacement.

DETAILED DESCRIPTION:
Patients with Tetralogy of Fallot have various degrees and levels of right ventricular outflow tract obstruction. They undergo surgical removal of the obstructing structures, which includes the pulmonary valve. The repair of the outflow tract is done utilizing a transannular patch. This approach, which is considered the standard of care, results in free pulmonary insufficiency, which may become severe and lead to right heart overloading and subsequent dilatation and dysfunction. This chronic overloading results in progressive tricuspid insufficiency and a suspected decline in effective pulmonary blood flow, cardiac output and right ventricle functional capabilities. Many patients develop progressive exercise intolerance, arrhythmias and severe cardiomegaly leading to dilated cardiomyopathy. The progressive decline in patient clinical status results in recommendations of pulmonary valve replacement to interrupt further dysfunction of the ventricles. Clinical improvement is generally seen among the patients and cardiac function is measurably improved in many cases, however the timing of surgery remains undefined and its impact on function improvement and recovery post -valve replacement is under serious debate and continuous discussion.

Preliminary work suggests that Magnetic Resonance Imaging (MRI) determined right to left ventricular volume ratio's of greater than 2:1 with associated tricuspid regurgitation, right ventricular regurgitant volumes of greater than 50%, and right ventricular ejection fractions less than 45% are common among patients with severe right ventricular failure and dysfunction. These patients are in need of pulmonary valve replacement and have routinely been referred for surgical intervention.

Patients with Aortic Coarctation have a localized malformation characterized by deformity of the aortic media, causing narrowing, usually severe, of the lumen of the vessel. Surgical repair or removal of this malformation is the treatment of choice however; the use of MRI to better determine the extent of damage or malformation would allow the surgeon to plan an operative strategy prior to opening the chest.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of Tetralogy of Fallot or Aortic Coarctation being Treated at Children's Healthcare of Atlanta at Egleston.

Exclusion Criteria:

* Those patients who do not meet the inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population is Patients with the diagnosis of Tetralogy of Fallot or Aortic Coarctation being Treated at Children's Healthcare of Atlanta at Egleston
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2002-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
(1) Determine Right and left ventricular volumes during all phases of the cardiac cycle. | 7 years
  (1) Determine Right and left ventricular volumes during all phases of the cardiac cycle.

CONTACTS AND LOCATIONS:
Overall Officials: James Parks, MD, Principal Investigator — Children's Healthcare of Atlanta, Sibley Heart Center Cardiology
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States